CLINICAL TRIAL: NCT06794099
Title: Applicability of CCR Assessment Criteria in PMMR Rectal Cancer Patients Treated with Neoadjuvant Chemoradiotherapy Combined with Immunotherapy
Brief Title: Study on the Applicability of CCR Criteria in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RECTUMCCR
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: PMMR/MSS Adenocarcinoma of the Colon or Rectum; Neoadjuvant Chemoradiotherapy; Immunotherapy; Complete Response
MeSH Terms: conditions — Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — This retrospective study does not involve biological specimens from patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NACRT Group: Participants in the neoadjuvant chemoradiotherapy (NACRT) group will receive standard neoadjuvant chemoradiotherapy. This typically involves a combination of chemotherapy drugs administered concurrently with radiation therapy targeted at the rectal tumor. The chemotherapy regimen may include drugs such as fluorouracil (5-FU) and leucovorin, or capecitabine, which are commonly used in the treatment of rectal cancer.
- NAICRT Group: Participants in the neoadjuvant chemoradiotherapy combined with immunotherapy (nICRT) group will undergo neoadjuvant chemoradiotherapy combined with immunotherapy. In addition to the standard chemotherapy and radiation therapy as described for the nCRT group, patients in this group will also receive immune checkpoint inhibitors (ICIs).

SUMMARY:
This study aims to explore how well the usual ways of checking if rectal cancer patients are free of disease signs after treatment work for a new treatment method. The new method combines chemotherapy, radiation, and immune-boosting drugs before surgery. We know these usual ways work for the standard treatment, but we're not sure if they're good enough for this new combo treatment. We'll look at patients with a specific type of rectal cancer that doesn't respond well to just immune-boosting drugs alone. By comparing how patients treated with the new method and the old method respond, we hope to find better ways to tell if the treatment is really working, which could help improve treatment plans for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. histopathologically confirmed adenocarcinoma;
2. pMMR/MSS tumors;
3. clinical staging of T3-T4 or any lymph node-positive T (N+);
4. no evidence of distant metastasis based on radiological examinations;
5. treatment with long-course chemoradiotherapy (LCRT) with or without immune checkpoint inhibitors (ICI);
6. post-neoadjuvant therapy evaluation with endoscopy and pelvic MRI.

Exclusion Criteria:

1. Presence of other active malignancies;
2. Having severe comorbidities, such as heart failure, severe hepatic or renal insufficiency, etc;
3. Lack of imaging and endoscopic examinations;
4. Treatment plan does not meet the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study evaluated medical records, endoscopic findings, and MRI images of rectal cancer patients who underwent neoadjuvant chemoradiotherapy (with or without immunotherapy) followed by surgery at Peking University Cancer Hospital between January 2019 and October 2024.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity, accuracy, and AUC | January 2025
  To evaluate the performance of clinical complete response (cCR) assessment criteria in patients treated with neoadjuvant chemoradiotherapy (nCRT) and neoadjuvant immunochemoradiotherapy (nICRT), we will utilize the area under the curve (AUC), accuracy, sensitivity, and specificity as key performance indicators. These metrics will help us assess the effectiveness of the cCR assessment criteria in both treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No